CLINICAL TRIAL: NCT01764854
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Parallel Design Study to Evaluate the Pharmacodynamics, Safety, and Tolerability of AZD1722 in End-Stage Renal Disease Patients on Hemodialysis
Brief Title: Pharmacodynamic Study of AZD1722 in End-stage Renal Disease Patients on Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardelyx (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5611C00001
Record Dates: First submitted 2013-01-04; First posted 2013-01-10 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: End Stage Renal Disease; Chronic Kidney Disease Stage 5; ESRD
Keywords: Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AZD1722- in patient (Experimental): Tenapanor administered in a clinical pharmacology unit
  Interventions: Drug: AZD1722 (in-patient)
- Placebo- in patient (Placebo Comparator): Placebo (size and color matched to experimental drug) administered in a clinical pharmacology unit
  Interventions: Drug: Placebo (in-patient)
- AZD1722 out-patient (Experimental): Tenapanor
  Interventions: Drug: AZD1722 (out-patient)
- Placebo out-patient (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1722 (in-patient) — doses between 5 and 60 mg BID may be administered based on tolerability in a CPU setting
  Other Names: RDX5791; Tenapanor
  Arms: AZD1722- in patient
Drug: Placebo (in-patient) — Placebo, size and color matched to experimental drug administered in a CPU
  Arms: Placebo- in patient
Drug: AZD1722 (out-patient) — doses between 5 and 45 mg BID
  Other Names: Tenapanor
  Arms: AZD1722 out-patient
Drug: Placebo — Placebo, size and color matched to experimental drug
  Arms: Placebo out-patient

SUMMARY:
The purpose of this study is to determine if the study drug is safe, tolerable and active in reducing fluid overload/weight gain between dialysis sessions for patients with End Stage Renal Disease on Hemodialysis.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacodynamics of the study drug in male and female patients with end-stage renal disease on hemodialysis. The study consists of a 2 week treatment-free run-in period where entry criteria are verified, a 4-week treatment period, of which the first week of treatment will be performed as an in-patient study in a clinical pharmacology unit (CPU) and the remaining three weeks of treatment will performed as an out-patient study, and a 2-week treatment-free follow-up period.

Safety assessments will be performed at regular intervals and will include clinical and vital signs, clinical laboratory evaluations, ECGs, and AE monitoring. Pharmacodynamic assessments will include, but are not limited to, interdialytic weight gain (IDWG), blood pressure, and stool sodium excretion. Pharmacokinetic assessments will include blood sampling for measurement of study drug plasma concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 80 years, inclusive;
* Body mass index between 18 and 45 kg/m2, inclusive;
* Ambulatory (≥ 6 months) maintenance hemodialysis;
* Stable dialysis treatment regimen 3x/week for ≥ 2 months prior to screening visit.

Exclusion Criteria:

* Currently taking diuretic medication;
* Has a urine production of ≥ 200 ml/day (based on a 24-hour measurement starting on Day -1 and completed prior to randomization);
* Predialysis systolic BP >200 mmHg or diastolic BP >110 mmHg on two successive occasions during the 2-week run-in period;
* Predialysis SBP < 110 mmHg on two successive occasions during the 2-week run-in period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, PhD, Study Director — Ardelyx, Inc.
Locations (3):
- United States (3):
  - Southwest Clinical Research Institute, Tempe, Arizona
  - Denver Nephrology, Denver, Colorado
  - DaVita Clinical Research, Minneapolis, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZD1722- in Patient | Placebo- in Patient | AZD1722 Out-patient | Placebo Out-patient
Started | 8 | 8 | 37 | 35
Completed | 8 | 8 | 31 | 33
Not Completed | 0 | 0 | 6 | 2
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — relocation | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1722- in Patient | Placebo- in Patient | AZD1722 Out-patient | Placebo Out-patient | Total
Number analyzed (Participants) | 8 | 8 | 37 | 35 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (8.3) | 54.4 (6.5) | 51.5 (11.5) | 49.3 (11.8) | 50.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 13 | 15 | 33
  Male | 6 | 5 | 24 | 20 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 13 | 10 | 24
  Not Hispanic or Latino | 7 | 8 | 24 | 25 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 14 | 19 | 45
  White | 2 | 2 | 18 | 16 | 38
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: centimeters] | 172.89 (9.31) | 172.05 (16.48) | 170.23 (10.80) | 170.20 (10.39) | 170.63 (10.84)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Weekly Interdialytic Weight Gain (IDWG)
Description: Patients are weighed pre dialysis prior to their first dialysis of the week. This measure looks at the change in pre-dialysis weight over time
Time Frame: Run-in period (Weeks -2 and -1) versus Week 4 (end of treatment)
Population: The out-patient arms were the only groups that were pre-specified to be included in this analysis since the in-patient arms were only treated for one week.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | AZD1722 Out-patient | Placebo Out-patient
Number analyzed (Participants) | 37 | 35
kilograms | -0.26 (0.939) | -0.23 (0.871)
Statistical Analysis 1: Comparison: AZD1722 Out-patient vs Placebo Out-patient; AZD1722 in-patient and Placebo in-patient are not included in this analysis since it was only a one week evaluation period and an effect was not expected. Also the size (n=8) of the group was too small to .perform this analysis; Test type: Superiority; p = 0.46, ANCOVA

2. Secondary Outcome: Stool Sodium Content
Description: The amount of sodium in a days worth of stool output
Time Frame: Days 1 through 7
Population: The in-patient arms were the only groups pre-specified to be used in this analysis since stool could only be collected in the clinical pharmacology unit (in-patient).
Measure: Mean (Standard Deviation); unit: mEq/day
Arm/Group | AZD1722- in Patient | Placebo- in Patient
Number analyzed (Participants) | 8 | 8
mEq/day | 36.62 (21.809) | 2.82 (2.655)
Statistical Analysis 1: Comparison: AZD1722- in Patient vs Placebo- in Patient; AZD1722 out-patient and Placebo out-patient were not included in this analysis since stool was only collected in the clinical pharmacology unit of the in-patient groups; Test type: Superiority; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: one month
Arm/Group | AZD1722- in Patient | Placebo- in Patient | AZD1722 Out-patient | Placebo Out-patient
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/37 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/8 | 3/8 | 2/37 | 1/35
Other Adverse Events (participants affected / at risk) | 6/8 | 2/8 | 3/37 | 21/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1722- in Patient (N=8) | Placebo- in Patient (N=8) | AZD1722 Out-patient (N=37) | Placebo Out-patient (N=35)
Syncope (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
local swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1722- in Patient (N=8) | Placebo- in Patient (N=8) | AZD1722 Out-patient (N=37) | Placebo Out-patient (N=35)
diarrhea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 3 (3) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days